CLINICAL TRIAL: NCT07348536
Title: Impact of Expanded Hemodialysis Prescription on Global Uremic Toxin Removal Compared With High-Volume Online Hemodiafiltration: A Randomized Open-Label Crossover Study
Brief Title: Expanded Hemodialysis Versus High-Volume Online Hemodiafiltration for Uremic Toxin Removal
Acronym: REMOV-HDx
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Olynka Vega, Principal investigator, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NMM-4853
Record Dates: First submitted 2025-12-22; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: End Stage Renal Disease (ESRD); Chronic Kidney Disease on Hemodialysis; Renal Dialysis; Uremia; Chronic; Hemodialysis; Hemodiafiltration
Keywords: Expanded hemodialysis; High-volume online hemodiafiltration; Medium cut-off dialysis membranes; Uremic toxin removal; Middle molecule clearance; Chronic kidney failure; Dialysis dose optimization; Dialysis treatment time; Global removal score
MeSH Terms: conditions — Kidney Failure, Chronic; Uremia; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Expanded Hemodialysis Prescriptions and High-Volume Online Hemodiafiltration (Experimental): Participants will receive three expanded hemodialysis sessions with different treatment durations (180, 210, and 240 minutes) in randomized order, followed by one session of high-volume online hemodiafiltration. Blood samples will be collected before and after each session to assess uremic toxin removal.
  Interventions: Device: Expanded Hemodialysis With Medium Cut-Off Membrane; Device: High-Volume Online Hemodiafiltration

INTERVENTIONS:
Device: Expanded Hemodialysis With Medium Cut-Off Membrane — Expanded hemodialysis will be performed using a medium cut-off dialysis membrane designed to enhance the removal of medium-sized uremic toxins while preserving albumin. Treatments will be delivered during regularly scheduled dialysis sessions with fixed dialysate flow and the maximum blood flow tolerated by the participant. Each participant will receive expanded hemodialysis sessions with three different treatment durations (180, 210, and 240 minutes), administered in randomized order following the long interdialytic interval. Blood samples will be collected before and after each session to assess removal of small and medium-sized uremic toxins.
  Other Names: Expanded hemodialysis; Medium cut-off hemodialysis
Device: High-Volume Online Hemodiafiltration — High-volume online hemodiafiltration will be delivered using post-dilution substitution during a standard dialysis session. Treatment will target a predefined convective volume consistent with high-volume hemodiafiltration while maintaining standard dialysis safety parameters. This intervention will be administered once to each participant after completion of the expanded hemodialysis sessions. Blood samples will be collected before and after the session to measure removal of small and medium-sized uremic toxins for comparison with expanded hemodialysis.
  Other Names: Online hemodiafiltration; High-volume hemodiafiltration; Post-dilution online hemodiafiltration

SUMMARY:
People with advanced kidney disease need dialysis to remove waste products from the blood. Some of these waste products, called uremic toxins, are small, while others are medium-sized and more difficult to remove. Poor removal of these toxins may contribute to symptoms and long-term complications in patients on dialysis.

Two dialysis techniques are commonly used to improve toxin removal beyond standard hemodialysis: expanded hemodialysis (HDx) using medium cut-off membranes, and high-volume online hemodiafiltration (HV-OL-HDF). Although both techniques are effective, the best way to prescribe expanded hemodialysis-particularly the ideal treatment time-has not been clearly defined.

The purpose of this study is to compare how well different treatment times of expanded hemodialysis remove small and medium-sized uremic toxins, and to compare these results with high-volume online hemodiafiltration. Toxin removal will be evaluated using a combined measurement called the Global Removal Score, which summarizes the removal of several important waste substances.

This is a single-center, randomized, open-label, crossover study. Adults receiving maintenance hemodialysis will receive three different expanded hemodialysis sessions with different treatment durations (180, 210, and 240 minutes), followed by one session of high-volume online hemodiafiltration. Blood samples will be taken before and after each dialysis session to measure toxin levels.

The results of this study may help determine whether expanded hemodialysis with shorter or standard treatment times can achieve toxin removal similar to high-volume hemodiafiltration, which could support more personalized and practical dialysis prescriptions.

DETAILED DESCRIPTION:
Expanded hemodialysis (HDx) using medium cut-off (MCO) membranes has been developed to improve the removal of medium-sized uremic toxins while maintaining effective clearance of small solutes. These medium-sized molecules have been associated with inflammation, cardiovascular disease, and other complications in patients with end-stage kidney disease. High-volume online hemodiafiltration (HV-OL-HDF) is currently considered a reference therapy for enhanced removal of these toxins, but its use may be limited by technical requirements, vascular access constraints, or resource availability.

While expanded hemodialysis has shown removal efficiency comparable to high-volume hemodiafiltration in prior studies, the optimal prescription of HDx-particularly the appropriate treatment duration-has not been clearly established. In routine clinical practice, dialysis dose is commonly guided by small-solute clearance (such as urea), which may not fully reflect the removal of medium-sized uremic toxins. A more comprehensive evaluation of toxin removal may help optimize dialysis prescriptions and improve treatment personalization.

This study is designed to compare the efficiency of uremic toxin removal across different expanded hemodialysis treatment durations and to contrast these results with high-volume online hemodiafiltration. Removal efficiency will be assessed using the Global Removal Score, a composite measure that integrates the removal rates of several small and medium-sized molecules while accounting for albumin loss.

The study is a single-center, randomized, open-label, crossover trial conducted in adult patients receiving maintenance hemodialysis. Each participant will receive three expanded hemodialysis sessions with different treatment durations (180, 210, and 240 minutes), administered in randomized sequences following the long interdialytic interval. After completion of the three expanded hemodialysis sessions, all participants will undergo one session of high-volume online hemodiafiltration with a predefined convective volume target.

During each study session, blood samples will be collected immediately before and after dialysis to measure concentrations of selected uremic toxins, including small solutes and medium-sized molecules. These measurements will be used to calculate individual and global removal rates for each dialysis modality and treatment duration. Standard dialysis parameters will be maintained according to institutional practice to ensure patient safety and consistency across sessions.

The crossover design allows each participant to serve as their own control, reducing variability related to patient-specific factors. The primary analysis will compare global toxin removal between expanded hemodialysis prescriptions and high-volume online hemodiafiltration, as well as across different HDx treatment durations.

The findings of this study may help clarify whether expanded hemodialysis with shorter or standard treatment times can achieve toxin removal comparable to high-volume hemodiafiltration. This information could support more individualized dialysis prescriptions and inform clinical decision-making in settings where high-volume hemodiafiltration is not feasible or routinely available.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* End stage renal disease Receiving maintenance hemodialysis three times per week on expanded hemodialysis as part of routine care for at least 1 month
* On dialysis treatment for more than 3 months
* Minimal or no residual urine output (less than 100 mL per day)
* Able and willing to provide written informed consent

Exclusion Criteria:

* Vascular access unable to support a blood flow of at least 300 mL/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-08-10 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2026-01-20 (Estimated)

PRIMARY OUTCOMES:
Global Removal Score of Uremic Toxins | During each dialysis intervention session (pre- and post-dialysis measurements), over a 4-week study period
  The Global Removal Score is a composite measure of dialysis efficiency that summarizes the percentage reduction of selected small and medium-sized uremic toxins during a dialysis session. It is calculated using the reduction ratios of urea, beta-2 microglobulin, myoglobin, prolactin, alpha-1 microglobulin, and alpha-1 acid glycoprotein, adjusted for albumin loss. Higher values indicate greater overall uremic toxin removal.

SECONDARY OUTCOMES:
Removal Rate of Individual Medium-Sized Uremic Toxins | During each dialysis intervention session (pre- and post-dialysis measurements), over a 4-week study period
  Percentage reduction of individual medium-sized uremic toxins, including beta-2 microglobulin, myoglobin, prolactin, alpha-1 microglobulin, and alpha-1 acid glycoprotein, measured before and after each dialysis session.
Removal Rate of Small Solutes | During each dialysis intervention session (pre- and post-dialysis measurements), over a 4-week study period
  Percentage reduction of small solutes, including urea and creatinine, measured before and after each dialysis session to assess small-molecule clearance across dialysis modalities and treatment durations.
Beta-2 Microglobulin Clearance by Kt/V | During each dialysis intervention session, over a 4-week study period
  Dialysis dose for beta-2 microglobulin expressed as Kt/V, calculated for each dialysis session to compare the kinetics of beta-2 microglobulin removal across expanded hemodialysis prescriptions and high-volume online hemodiafiltration.

CONTACTS AND LOCATIONS:
Overall Officials: Olynka Vega, MS, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutrición Salvador Zubirán
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubiran, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared publicly. This study involves a small, single-center cohort with detailed clinical and laboratory data, and sharing individual-level data could increase the risk of participant re-identification. In addition, the data are collected for a specific mechanistic research purpose and are not intended for secondary analyses outside the scope of the approved protocol. Aggregate results will be reported through scientific publications and presentations.